CLINICAL TRIAL: NCT01820299
Title: Phase I Assay-guided Trial of Anti-inflammatory Phytochemicals in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael Lilly, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101839
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Solid Cancers
MeSH Terms: interventions — Grape Seed Extract; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Grape Seed Extract and Vitamin D (Experimental): All patients will take Grape Seed Extract from Day 1 to Day 21. All patients will take Grape Seed Extract and Vitamin D together from Day 22 until Day 64. For all patients on the study, patients will take Vitamin D once a day at a dose of 4000IU.
  Interventions: Drug: Grape Seed Extract; Drug: Vitamin D

INTERVENTIONS:
Drug: Grape Seed Extract — All patients enrolled to the study will take Grape Seed Extract alone for 21 days.
  Other Names: GSE
Drug: Vitamin D — From Day 22 until Day 64 of the study, patients will take Grape Seed Extract and Vitamin D together. Patients will take Vitamin D once at a day at 4000 IU.

SUMMARY:
This study is for subjects with solid cancers (gastrointestinal, lung, breast, prostate, lymphoma or cancer of the lymph nodes). The overall goal of this study is to identify plant-derived phytochemicals that can safely reduce systemic inflammation (inflammation throughout the entire body) in subjects with advanced cancer.

DETAILED DESCRIPTION:
This study will look at oligomeric procyanidin complex (OPC) and vitamin D3. OPC is the major part of Grape Seed Extract (GSE). Researchers are in looking at the combination of GSE and vitamin D in subjects with solid cancers (gastrointestinal, lung, breast, prostate, lymphoma or cancer of the lymph nodes). Researchers will examine the safety of the GSE and vitamin D when GSE is given at different doses. Researchers will also look at the effects of GSE and vitamin D on your quality of life and your body. In particular, they will look at differences in biomarkers in your blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histological diagnosis of cancer
* Subjects must be 21 or more years of age
* Subjects must have metastatic or locally advanced, unresectable cancer. Cancer must be "active" (i.e. demonstrable by physical examination, blood tests, or radiographical procedures).
* Subjects may not initiate a new form of cancer therapy, non-steroidal or steroid anti-inflammatory agents, or antibiotics during the study period or for 4 weeks prior to the start of study agents.
* Subjects must be able to give written consent to the study.
* Subjects must have adequate hematologic, renal, and hepatic function at baseline, as follows:
* Hematology parameters: ANC >1500/mcL, platelets > 100,000/mcL, Hgb >8.0gm/dL
* Renal Function: Creatinine <1.8mg/mL
* Liver Function: Total bilirubin ≤ULN, AST and ALT <1.5xULN, Alk phosphatase <2.5xULN
* Subjects must have normal serum phosphate and serum calcium levels:
* Serum Phosphate > 2.3 and < 4.8 mg/dL
* Serum Calcium > 8.5 and < 10.5
* Subjects may be receiving anti-cancer treatment, but this treatment should be have been instituted at least 4 weeks prior to enrollment, and may not change during the study period.

Exclusion Criteria:

* Uncontrolled cancer requiring the institution of new anti-cancer therapy during the study period.
* Presence of any severe or uncontrolled concurrent medical condition which, in the opinion of the investigator, would increase the risk of serious toxicity from the study drugs.
* Any uncontrolled systemic inflammatory disease or infection requiring antibiotics, non-steroidal, or steroidal anti-inflammatory agents.
* Initiation of strong antioxidant supplements during treatment, or ongoing use of supplements containing concentrated plant-derived polyphenols (pine bark, grape seed, green tea, milk thistle extracts; resveratrol; ellagic acid)
* Pregnancy or breast feeding
* Any history of allergies to grapes or grape seed.
* Current treatment with lenalidomide, thalidomide, imipquimod, interferon, cytokines (G-CSF, GM-CSF, IL-1Rα), TNFα antagonists, or Lithium.
* History of sarcoidosis
* History of hypercalcemia
* Use of any non-protocol vitamin D supplementation.
* Uncontrolled hypertension
* Current treatment with warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximally-tolerated dose of Grape Seed Extract in Patients with Solid Tumors | 2 years
  Decisions to escalate or expand a dose level will be based only on the GSE-only treatment period (day 1-21). To be evaluable for toxicity, a patient must receive at least 3 weeks of GSE treatment, or have experienced dose-limiting toxicity (DLT). All patients enrolled are to be fully followed for toxicity, but any patients who are not evaluable for toxicity will be replaced.

SECONDARY OUTCOMES:
IL6 Response | 2 years
  Plasma IL-6 levels before and after 21 days and 63 days of GSE treatment will be quantified to estimate the dose response relationship between GSE dose and reduction in inflammation.

OTHER OUTCOMES:
Measurement of Other Inflammatory Markers | 2 years
  Other markers that will be measured will include serum CRP, albumin, AGEs (advanced glycation end products), rAGE (soluble receptor for AGEs), 25-OH-vitamin D3, and urine for oxidative damage DNA biomarkers (urinary 8-oxoGua and 8-oxodG). Correlations between dose and change in these parameters from before to 21, 63 days after start of GSE dosing will be described.
Quality of Life Questionnaires | 2 years
  Serial QOL assessments will be made by the FACT series of QOL questionnaires
Effect of Vitamin D3 on Anti-Inflammatory Effects of GSE | 2 years
  The ability of a fixed dose of vitamin D3 (4000 IU daily) to further suppress IL-6 levels in subjects on GSE treatment will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States